CLINICAL TRIAL: NCT00629343
Title: A Phase I Dose-Escalation Study Of Azacitidine In Combination With Temozolomide In Patients With Unresectable Or Metastatic Soft Tissue Sarcoma or Malignant Mesothelioma
Brief Title: Phase I Dose-Escalation Study Of Azacitidine In Combination With Temozolomide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Schering-Plough (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC3255
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Soft Tissue Sarcoma; Mesothelioma
Keywords: Soft Tissue Sarcoma; Mesothelioma; Azacitidine; Temozolomide; Temodar
MeSH Terms: conditions — Sarcoma; Mesothelioma | interventions — Azacitidine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Subjects will receive azacitidine in combination with temozolomide
  Interventions: Drug: Azacitidine; Drug: Temozolomide

INTERVENTIONS:
Drug: Azacitidine — Azacitidine will be delivered sub-cutaneously for 5 days
  Other Names: Vidaza
Drug: Temozolomide — Temozolomide will be given starting on day 8 for 5 days at a dose of 200 mg/m2 po qd x 5 days
  Other Names: Temodar

SUMMARY:
The purpose of this study is to determine safety and toxicity for the combination of Temozolomide and Azacitidine in the treatment of Advanced Soft Tissue Sarcoma or Malignant Mesothelioma. This is a single-center, open-label, single-arm Phase I dose-escalation trial. Patients will be evaluated with complete history and physical as well as laboratory studies (complete blood count, metabolic panel, liver function tests), biopsy, and imaging of all sites of measurable disease. This study will be conducted over the course of 3 years.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the clinical and laboratory toxicities as well as acceptability/tolerance of this dose schedule of combined drug treatment with temozolomide and azacitidine.

Secondary objectives include determination of biochemical response to azacitidine as defined as change in methylation status. The investigators will specifically be looking at changes in genome wide methylation patterns as determined by two high-throughput platforms:

1. A single nucleotide polymorphism chip-based method (MSNP) for genome wide epigenetic profiling
2. CpG island promoter arrays will be performed to focus on promoter methylation status.

The investigators will also monitor clinical response, time to progression and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed soft tissue sarcoma or mesothelioma.
* Ineligible for other high priority national or institutional study.
* Non-pregnant, non-lactating.
* Recurrent or progressive disease defined as an increase in size of any existing tumor mass, or the development of new tumor mass or masses, which is not amenable to definitive surgical therapy.
* Measurable disease defined as lesions that can be measured in at least one dimension by physical examination or by means of medical imaging techniques. Ascites and pleural effusions will not be considered measurable disease.
* Prior chemotherapy is allowed with the exception of prior treatment with Temozolomide or Azacitidine. Patients must have received prior 1st line therapy. There is no upper limit to the number of prior therapies received. Prior treatment with an alkylating agent is acceptable.
* Prior radiation therapy is allowed.
* At least 4 weeks since prior chemotherapy or at least 6 weeks since prior radiation therapy.
* Patients may have had another cancer but there must be convincing clinical evidence that the sarcoma is the disease requiring therapeutic intervention. (i.e. Several sarcoma patients have had had a prior cancer [Hodgkin's disease or breast cancer] treated years previously and then developed a clinically active sarcoma.)
* Clinical parameters: Life expectancy > 3 months, Age > 18 years, Performance Karnofsky performance status of greater than or equal to 60%.
* Required initial laboratory data:

  * Absolute neutrophil count > 1,500/mm3
  * Hemoglobin > 10.0 g/dl
  * Platelet count > 100,000/mm3
  * Total Bilirubin < 1.5 times upper limit of normal (ULN) for the laboratory.
  * Transaminases: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels must be < 2 x ULN. If there is known hepatic metastasis, transaminases may be < 5 times upper limit of normal.
  * Serum creatinine levels < 1.5 x ULN.
  * Women of child-bearing potential must have a negative serum pregnancy test prior to initiation of treatment.
* Men and women of child-bearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter (approximately 3 months).
* Capable of providing written, informed consent. Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks and discomforts.
* No serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g. serious infection).
* No uncontrolled central nervous system metastases.

Exclusion Criteria:

* Known or suspected hypersensitivity to azacitidine or mannitol
* Pregnant or breast-feeding
* Histology other than soft-tissue sarcoma or mesothelioma
* Active or uncontrolled infection or other serious systemic disease
* Prior treatment with temozolomide or azacitidine
* Pregnant or lactating women
* Uncontrolled central nervous system metastases
* Liver metastases
* Patients will not be excluded if they do not wish to participate in the second biopsy for tissue evaluation
* Subjects who have not had prior chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N Taub, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants signed a consent form and four were determined to be ineligible, resulting in 23 assigned to treatment.
Groups:
- Azacitidine 25mg: Cohort 1: Participants received 25 mg Azacitidine sub-cutaneously, and 200 mg/m2 Temozolomide orally; both once a day on Days 1 - 5 of a 28-day cycle.
- Azacitidine 50 mg: Cohort 2: Participants received 50 mg Azacitidine sub-cutaneously, and 200 mg/m^2 Temozolomide orally; both once a day on Days 1 - 5 of a 28-day cycle.
- Azacitidine 75 mg: Cohort 3: Participants received 75 mg Azacitidine sub-cutaneously, and 200 mg/m^2 Temozolomide orally; both once a day on Days 1 - 5 of a 28-day cycle.
Period: Dose Level 1: Azacitidine 25mg
Arm/Group | Azacitidine 25mg | Azacitidine 50 mg | Azacitidine 75 mg
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Dose Level 2: Azacitidine 50 mg
Arm/Group | Azacitidine 25mg | Azacitidine 50 mg | Azacitidine 75 mg
Started | 0 | 3 | 0
Completed | 0 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Dose Level 3: Azacitidine 75mg
Arm/Group | Azacitidine 25mg | Azacitidine 50 mg | Azacitidine 75 mg
Started | 0 | 0 | 17
Completed | 0 | 0 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Azacitidine 25 mg: Cohort 1: Participants received 25 mg Azacitidine sub-cutaneously, and 200 mg/m^2 Temozolomide orally; both once a day on Days 1 - 5 of a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Azacitidine 25 mg | Azacitidine 50 mg | Azacitidine 75 mg | Total
Number analyzed (Participants) | 3 | 3 | 17 | 23
Age, Customized [Count of Participants; unit: Participants]
  ≥ 18 years | 3 | 3 | 17 | 23
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 0 | 0 | 0 | 0
  Unknown | 3 | 3 | 17 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Temozolomide
Description: Maximum tolerated dose of temozolomide when used in combination with azacitidine
Time Frame: Up to 26 weeks for each dosing cohort
Measure: Number; unit: mg/m^2
Arm/Group | Treatment
Number analyzed (Participants) | 23
mg/m^2 | 200

2. Primary Outcome: Maximum Tolerated Dose of Azacitidine
Description: Maximum tolerated dose of azacitidine when used in combination with temozolomide
Time Frame: Up to 26 weeks for each dosing cohort
Measure: Number; unit: mg/m^2
Arm/Group | Treatment
Number analyzed (Participants) | 23
mg/m^2 | 75

ADVERSE EVENTS:
Time Frame: up to 59 months after enrollment
Arm/Group | Azacitidine 25 mg | Azacitidine 50 mg | Azacitidine 75 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 15/17
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 15/17
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine 25 mg (N=3) | Azacitidine 50 mg (N=3) | Azacitidine 75 mg (N=17)
Death due to progression of disease (General disorders) | 0 | 0 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes